CLINICAL TRIAL: NCT04974346
Title: Para-aortic Prophylactic Irradiation for Locally Advanced Cervical Cancer: a Prospective, Randomized, Multicenter Study
Brief Title: Para-aortic Prophylactic Irradiation for Locally Advanced Cervical Cancer
Acronym: PAILACC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CARTOnG 2101
Record Dates: First submitted 2021-07-04; First posted 2021-07-23 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2021-07

CONDITIONS: Cervical Cancer
Keywords: locally advanced cervical cancer; para-aortic radiotherapy; concurrent radiochemotherapy; PET-CT
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study arm (Experimental): External beam radiotherapy:
  Pelvic and para-aortic radiotherapy 45-50.4Gy/25-28 fractions. PET-CT positive lymph node should be boost to a dose of 60Gy or higher. Parametrium(both) should be boost to a dose from 50Gy to 60Gy.
  Concurrent chemotherapy:
  Weekly cisplatin 40mg/m2 during external beam radiotherapy.
  Brachytherapy:
  High dose rate(HDR) Brachytherapy. The dose of high-risk clinical target volume(HR CTV) D90 or Point A should be 85Gy+/-10%. The dose of intermediate-risk clinical target volume(IR CTV) D98 should be 60Gy at least.
  Interventions: Radiation: Paraaortic prophylactic irradiation and pelvic definitive concurrent chemoradiation
- control arm (Active Comparator): External beam radiotherapy:
  Pelvic radiotherapy 45-50.4Gy/25-28 fractions. PET-CT positive lymph node should be boost to a dose of 60Gy or higher. Parametrium(both) should be boost to a dose from 50Gy to 60Gy.
  Concurrent chemotherapy:
  Weekly cisplatin 40mg/m2 during external beam radiotherapy.
  Brachytherapy:
  HDR Brachytherapy. The dose of HR CTV D90 or Point A should be 85Gy+/-10%. The dose of IR CTV D98 should be 60Gy at least.
  Interventions: Radiation: Pelvic definitive concurrent chemoradiation

INTERVENTIONS:
Radiation: Paraaortic prophylactic irradiation and pelvic definitive concurrent chemoradiation — The para-aortic area, from left renal vein level to abdominal aorta bifurcation level，will be prophylactic irradiation. The other intervention is the same as control arm.
  Arms: study arm
Radiation: Pelvic definitive concurrent chemoradiation — Pelvic definitive concurrent chemoradiation, including external beam radiotherapy, concurrent chemotherapy and brachytherapy.
  Arms: control arm

SUMMARY:
Para-aortic lymph node metastasis is a poor prognostic factor for locally advanced cervical cancer, but false negative diagnosis is easy to occur. The aim of this trial was to investigate whether para-aortic prophylactic radiotherapy improves disease-free survival in patients with positive pelvic lymph nodes below the common iliac artery.

DETAILED DESCRIPTION:
This clinical trial enrolled participants with locally advanced cervical cancer with positive pelvic lymph nodes below the common iliac region diagnosed by Positron emission tomography-computed tomography(PET-CT). Participants should be able to receive concurrent cisplatin chemotherapy. No anti-tumor treatment was given before randomization. Participants will be randomly assigned to two groups. The study group will receive radiotherapy of pelvic and para-aorta, concurrent chemotherapy and brachytherapy, and the control group will receive pelvic radiotherapy, concurrent chemotherapy and brachytherapy.

ELIGIBILITY:
Inclusion Criteria:

* The patients voluntarily participated in the study and signed the informed consent
* 18-75 female
* Cervical squamous cell carcinoma / adenocarcinoma / adenosquamous cell carcinoma
* According to International Federation of Gynecology and Obstetrics(FIGO) 2009 stage, stage ⅠB2 - ⅣA with positive pelvic lymph nodes and negative common iliac and paraaortic lymph nodes diagnosed by PET-CT
* Cisplatin chemotherapy is acceptable
* Eastern Cooperative Oncology Group(ECOG) score 0-1
* The expected survival was more than 6 months
* Women of childbearing age must have a pregnancy test (serum or urine) within 7 days before enrollment, and the result is negative, and they are willing to use appropriate contraceptive methods during the test
* According to the judgment of the researcher, those who can comply with the trial protocol

Exclusion Criteria:

* Uncontrolled severe infection
* Combined with other malignant tumor patients who need treatment and / or new diagnosis within 5 years
* The patient has received anti-tumor treatment
* Liver cirrhosis, decompensated liver disease, chronic renal insufficiency and renal failure
* History of immunodeficiency, including HIV positive or other acquired congenital immunodeficiency disease
* Myocardial infarction, severe arrhythmia and grade 2 or more congestive heart failure (NYHA classification)
* Patients with previous pelvic artery embolization
* Previous radiotherapy for pelvic malignant tumor
* There was a history of severe allergic reaction to platinum containing chemotherapy drugs
* Complications, need to be taken during the treatment of liver and kidney function damage drugs, such as tuberculosis
* The patients who could not understand the content of the experiment and could not cooperate and refused to sign the informed consent
* Patients with accompanying diseases or other special circumstances that seriously endanger the safety of patients or affect the completion of the study

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 455 (Estimated)
Dates: Start 2021-08-02 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2030-08-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival rate | 3-year
  the percentage of participants in the group whose disease is likely to remain stable

SECONDARY OUTCOMES:
Overall survival rate | 3-year
  the percentage of participants in the group who survives
Para-aortic recurrence rate | 3-year
  the percentage of participants involved by recurrence in the area of para-aortic lymph node
Distant recurrence rate | 3-years
  the percentage of participants involved by recurrence in any organ or tissue except pelvic and para-aortic area
Side effects | 3-year
  side effects associated with treatment
Quality of life (QOL) assessed by EORTC QLQ-C30 v3 | 1-month and 6-month
  an individual's perception of their position in life in the context of the culture and value systems in which they live and in relation to their goals, expectations, standards and concerns (assessed by EORTC QLQ-C30 v3 )
Quality of life (QOL) assessed by EORTC QLQ-CX24 | 1-month and 6-month
  an individual's perception of their position in life in the context of the culture and value systems in which they live and in relation to their goals, expectations, standards and concerns (assessed by EORTC QLQ-CX24)

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou
  - Jinhua Municipal Central Hospital Medical Group, Jinhua
  - Lishui People's Hospital, Lishui
  - Ningbo First Hospital, Ningbo
  - Taizhou Central Hospiatl, Taizhou
  - Chongqing University Three Gorges Hospital, Wanzhou

IPD SHARING:
Plan to Share IPD: No